CLINICAL TRIAL: NCT03846700
Title: Non Inferiority Clinical Randomized Trial Comparing Disobstrucitve Power in Patients With LUTS by BHP (Evaluated With Invasive Advanced Urodynamic Tests) That Underwent to Aquablation, Holep and PVP
Brief Title: Urodynamic Evaluation of Disobstrucitve Power of Aquablation VS Laser Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bari (Other)
Collaborators: Gaetano de Rienzo (Unknown); Pasquale Ditonno (Unknown); Francesco Di Modugno (Unknown); Michele Battaglia (Unknown); Giuseppe Lucarelli (Unknown); Marco Spilotros (Unknown)
Responsible Party: Principal Investigator, Paolo Minafra, Resident Doctor, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2019-02-15; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Aquablation

STUDY DESIGN:
Intervention Model Description: non inferiority, blinded, prospective, randomized clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- aquablation (Experimental): patients with prostatic volume included between 30 and 120 ml will be treated with water jet (aquablation). patients with prostatic volume > 65 ml will be compared with holep arm and patients with prostatic volume included between 30 and 65 ml will be compared with pvp arm.
  Interventions: Device: aquablation
- holep (Active Comparator): patients with prostatic volume > 65 ml will be treated with holmium laser technique (Holep)
  Interventions: Device: holep
- pvp (Active Comparator): patients with prostatic volume included between 30 and 65 ml will be treated with photoselective vaporization of prostate (pvp).
  Interventions: Device: pvp

INTERVENTIONS:
Device: aquablation — minimally invasive, robot-assisted and ultrasound-guided ablation of the prostate in targeted way and in "heat-free" way working by high pression water jet
  Arms: aquablation
Device: holep — holmium laser enucleation of prostate
  Arms: holep
Device: pvp — photoselectivevaporization of prostate
  Arms: pvp

SUMMARY:
in the last decade, lots of attemps have been done to identify new technologies able to reply the efficacy of gold standard technique for treating BPH, but with a better safety profile. The introduction of laser techniques allowed to reduce complication rates. Among these, considerable importance had Holep and PVP. Aquablation is a recent technique for LUTS treatment. It is minimally invasive, robot-assisted and ultrasound-guided to ablate the prostate in targeted way and in "heat-free" way. It works with high pression water jet. However, in literature informations about disobstructive capacity of minimally invasive techniques, evaluated with invasive urodynamic tests, are low.

The enrolled subjects will undergo surgical treatment with one of the techniques under study: Aquablation, HoLEP or PVP.

Outpatient visits will be performed at 1, 3 and 6 months after the surgical treatment. During the sixth month visit an invasive urodynamic examination will be performed

DETAILED DESCRIPTION:
in the last decade, lots of attemps have been done to identify new technologies able to reply the efficacy of gold standard technique for treating BPH, but with a better safety profile. The introduction of laser techniques allowed to reduce complication rates. Among these, considerable importance had Holep and PVP. Aquablation is a recent technique for LUTS treatment. It is minimally invasive, robot-assisted and ultrasound-guided to ablate the prostate in targeted way and in "heat-free" way. It works with high pression water jet.

However, in literature informations about disobstructive capacity of minimally invasive techniques, evaluated with invasive urodynamic tests, are low.

In particular, about Aquablation, just in one trial is reported the reduction of BOOI, from 49 to 24 in 6 months after surgery, but this information is not associated with standard deviation and statistical significance.

Perreira-Carreia, J.A. et al, in 2012 reported a medium BOOI variation after 6 months by surgery, from 60 to 8,7 (p<0,001) even if procedure was conducted with laser 120 W.

In 2014 Know, O. and coll., reported BOOI reduction after Holep from 54,9 ± 30,2 to 3,4 ± 17,4 (p<0,001).

Actually, there are not trials comparing Aquablation with others mininvasive techniques to treat LUTS by BHP (in particular Holep and PVP).

This comparison is very interesting because of the specific benefits of each technique.

General and specific aims:

1. non inferiority evaluation of the BOOI variations in patients with LUTS caused by cervico-urethral obstruction by BHP undergone to endoscopic surgery with aquablation versus patients operated with laser endoscopic surgery (primary goal);
2. Evaluation of the IPSS score variations in two groups of patients,
3. Evaluation of Qmax variations with uroflowmetry and post-voiding residue in two groups;
4. Evaluation of sexual satisfaction by IIEF-5 survey and evaluation of presence of anejaculation in two groups;
5. Evaluation of total-PSA variation in two groups;
6. Evaluation of operative times, hospitalization and variations of haemoglobin and haematocrit value in two groups;
7. Evaluation of appearing of side effects (grade 1 and ≥ 2 by Clavien-Dindo) occurred in perioperative period and at 1, 3 and 6 months after surgery;

Inclusion criteria:

* age ≥ 40 years and <90 years;
* moderate-to-severe lower urinary tract symptoms (IPSS ≥ 12)
* poor efficacy or tolerance to medical therapy for BPH
* transrectal ultrasound prostate volume between 30 and 120 ml
* ability to express written informed consent.

Exclusion criteria:

* previous surgical treatments for BPH
* indwelling bladder catheter or clean intermittent catheterization
* bladder stones
* severe detrusor hypocontractility (BCI <50) or detrusorial acontractility
* urethral strictures
* neurological bladder
* not replaceable anticoagulant or antiplatelet drugs for severe cardiological comorbidity
* bladder cancer;
* diagnosis or clinical suspicion of prostatic cancer;

Treatment The enrolled subjects will undergo surgical treatment with one of the techniques under study: Aquablation, HoLEP or PVP.

The study population will be divided into two cohorts based on prostate volume measured by transrectal ultrasound. Thereafter, patients with a prostate volume between 30 and 65 ml will be assigned to the aquablation arm or PVP arm, while patients with a prostate volume over 65 ml will be subjected to aquablation or HoLEP. The assignment to each of the arms will be randomized, using an on-line software for block randomization.

Follow-up:

Follow-up visits will be conducted by a blinded research team. Outpatient visits will be performed at 1, 3 and 6 months after the surgical treatment. During the sixth month visit an invasive urodynamic examination will be performed with cystomanometry and pressure-flow study.

ELIGIBILITY:
Inclusion Criteria:

* moderate-to-severe lower urinary tract symptoms (IPSS ≥ 12)
* poor efficacy or tolerance to medical therapy for BPH
* transrectal ultrasound prostate volume between 30 and 120 ml
* ability to express written informed consent.

Exclusion Criteria:

* previous surgical treatments for BPH
* indwelling bladder catheter or clean intermittent catheterization
* bladder stones
* severe detrusor hypocontractility (BCI <50) or detrusorial acontractility
* urethral strictures
* neurological bladder
* not replaceable anticoagulant or antiplatelet drugs for severe cardiological comorbidity
* bladder cancer;
* diagnosis or clinical suspicion of prostatic cancer

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
BOOI variations | 6 months
  non inferiority evaluation of the BOOI variations in patients with LUTS caused by cervico-urethral obstruction by BHP undergone to endoscopic surgery with aquablation versus patients operated with laser endoscopic surgery

SECONDARY OUTCOMES:
IPSS score | 1, 3 and 6 months
  Evaluation of the IPSS score variations in two groups of patients,
Qmax | 1, 3 and 6 months
  Evaluation of Qmax variations with uroflowmetry and post-voiding residue in two groups;
sexual satisfaction | 1, 3 and 6 months
  Evaluation of sexual satisfaction by IIEF-5 survey and evaluation of presence of anejaculation in two groups;

OTHER OUTCOMES:
PSA | 1, 3 and 6 months
  Evaluation of total-PSA variation in two groups
complications | 1, 3 and 6 months
  Evaluation of appearing of side effects (grade 1 and ≥ 2 by Clavien-Dindo) occurred in perioperative period and at 1, 3 and 6 months after surgery;

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bari "Aldo Moro", Bari, Italy

IPD SHARING:
Plan to Share IPD: No